CLINICAL TRIAL: NCT00298506
Title: An Open, Prospective Study to Assess the Efficacy and Safety of FK506 Combined MMF in the Treatment of Class III，IV，V + IV or V + III Lupus Nephritis
Brief Title: Study to Assess the Efficacy and Safety of FK506 Combined With Mycophenolate Mofetil (MMF) in Lupus Nephritis (III/IV/V)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing University School of Medicine (Other)
Responsible Party: Principal Investigator, Zhi-Hong Liu, M.D., Research Institute of Nephrology, Nanjing University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NJCT-0601
Record Dates: First submitted 2006-03-01; First posted 2006-03-02 (Estimated); Last update posted 2011-09-29 (Estimated); Status verified 2011-09

CONDITIONS: Lupus Nephritis
Keywords: Tacrolimus; Mycophenolate mofetil; Cyclophosphamide; Lupus nephritis; Treatment
MeSH Terms: conditions — Lupus Nephritis | interventions — Tacrolimus; Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- FK506+MMF (Active Comparator)
  Interventions: Drug: Multitherapy

INTERVENTIONS:
Drug: Multitherapy — Tacrolimus,4mg/d, MMF 1.0g/d
  Other Names: FK506,Prograf,Tacrolimus; MMF,cellcept,mycophenolate mofetil

SUMMARY:
This is an open, prospective study to assess the efficacy and safety of Tacrolimus (FK506) combined with MMF in the treatment of class III, IV, V + IV or V + III lupus nephritis.

DETAILED DESCRIPTION:
1. To assess the efficacy of FK506 combined with MMF vs intravenous CTX pulses in treatment of class Ⅲ, Ⅳ, Ⅴ + Ⅳ or Ⅴ + Ⅲ LN.
2. To investigate the safety and tolerability of FK506 combined with MMF vs intravenous CTX pulses in the treatment of class Ⅲ, Ⅳ, Ⅴ + Ⅳ or Ⅴ + Ⅲ LN.
3. To explore the dosing of FK506 combined with MMF and their effective range of blood concentration.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients with a diagnosis of systemic lupus erythematosus (SLE) according to the criteria of American Rheumatic Association, 1982, aged between 12-50 years, with score of SLE-DAI (Disease Active Index) of more than 12 (not including class V LN).
2. Patients diagnosed according to ISN/RPS 2003 classification criteria: class Ⅲ, Ⅳ, Ⅳ + Ⅴ, Ⅲ + Ⅴ LN by renal biopsy within 3 months, CI< 4，Scr< 3 mg/dl.
3. Patients with a proteinuria ≥ 1.5 g/24h, or active urine sediment.
4. Patients who signed written informed consent forms (patients less than 18 years old with their parents/legal representative' signatures), and have given their consent to follow all study procedures and follow-ups.

Exclusion Criteria:

1. Patients who have received treatment of cytotoxic drugs such as cyclophosphamide (CTX), cyclosporine A for more than 1 week within three months.
2. Patients with serum creatinine ≥ 3 mg/dl（265 μmol/L).
3. Patients with severe infection or central nervous system symptoms.
4. Patients who have impaired liver function, with ALT/GPT or AST/GOT twice more than the normal upper limit or who have active hepatitis.
5. Patients who have abnormal blood glucose, with a fasting blood glucose > 6.2 mmol/L or post meal blood glucose > 11.2 mmol/L.
6. Patients who are pregnant or lactating.
7. Patients who are known to be allergic to a macrolide.

Ages: 12 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 120 (Actual)
Dates: Start 2005-09; Primary Completion 2008-12 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
To assess the efficacy of FK506 combined with MMF versus intravenous CTX pulses in treatment of LN | 18 months

SECONDARY OUTCOMES:
To investigate the safety and tolerability of FK506 combined with MMF versus intravenous CTX pulses | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Lei-Shi Li, M.D., Study Director — Research Institute of Nephrology, Jinling Hospital, Nanjing University School of Medicine
Locations (2):
- China (2):
  - Research Institute of Nephrology, Jinling Hospital, Nanjing University School of Medicine, Nanjing, Jiangsu
  - Research Institute of Nephrology, Jinling Hospital, Nanjing, Jiangsu

REFERENCES:
- [Derived] Bao H, Liu ZH, Xie HL, Hu WX, Zhang HT, Li LS. Successful treatment of class V+IV lupus nephritis with multitarget therapy. J Am Soc Nephrol. 2008 Oct;19(10):2001-10. doi: 10.1681/ASN.2007121272. Epub 2008 Jul 2. PMID 18596121